CLINICAL TRIAL: NCT04584580
Title: D-dimer Adjusted Versus Therapeutic Dose Low-molecular-weight Heparin in Patients With COVID-19 Pneumonia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ashraf M Madkour, Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FMASU P35/ 2020
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Coronavirus Disease (COVID)19
MeSH Terms: conditions — COVID-19 | interventions — Heparin, Low-Molecular-Weight; Enoxaparin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic dose low-molecular-weight heparin (LMWH) (Active Comparator): Therapeutic dose low-molecular-weight heparin from admission until the end of hospital stay Enoxaparin 1 mg/kg subcutaneous every 12 hours
  Interventions: Drug: low-molecular-weight heparin
- D-dimer levels and weight adjusted low-molecular-weight heparin (LMWH)therapy (Experimental): from admission until the end of hospital stay. Patients will be stratified according to their body weight and D-dimer level and receive LMWH
  D-Dimer level Body Weight LMWH dose
  <1 mg/dl <100kg Enoxaparin 40mg OD 100-150kg Enoxaparin 40mg BD >150kg Enoxaparin 60mg BD
  1-3 mg/ dl <100kg Enoxaparin 40mg BD 100-150kg Enoxaparin 80mg BD >150kg Enoxaparin 120mg BD
  >3 mg/ dl Enoxaparin 80mg BD
  Interventions: Drug: low-molecular-weight heparin

INTERVENTIONS:
Drug: low-molecular-weight heparin — low-molecular-weight heparin administered via subcutaneous injection
  Other Names: Enoxaparin

SUMMARY:
evaluation of the efficacy and safety of D-dimer adjusted heparin versus therapeutic dose heparin in patients with COVID-19 Pneumonia.

DETAILED DESCRIPTION:
The following will be done for enrolled patients:

1. Data collection: name, age, sex, special habits of medical importance (i.e. smoking, drug abuse), comorbid conditions.
2. Clinical examination Vital data Local chest examination
3. Measurement of oxygen saturation using pulse oximeter
4. Laboratory investigations:

   Complete blood count with differential count Liver and kidney functions D-dimer level Coagulation profile
5. Radiology work up ( Chest X-ray-High resolution computed tomography of the chest- computed tomography of the chest with pulmonary angiography as needed)
6. Sepsis-induced coagulopathy score (SIC score)
7. Sequential organ failure score (SOFA score)
8. Patients will receive treatment according to the hospital guidelines for different disease stratification severity

ELIGIBILITY:
Inclusion Criteria:

* All adult (>18 years) patients from both sexes with COVID-19 pneumonia with positive nucleic acid test for severe acute respiratory syndrome Coronavirus (SARS-CoV-2) hospitalized either in the ward or intensive care unit

Exclusion Criteria:

* Patients with absolute contraindication of pharmacological thromboprophylaxis and/ anticoagulation
* Congenital hemorrhagic disorders
* Hypersensitivity to heparin
* Personal history of heparin-induced thrombocytopenia
* Active major bleeding or conditions predisposing to major bleeding. Major bleeding is defined as fulfilling any one of these three criteria: a) occurs in a critical area or organ (e.g.intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, intra-uterine or intramuscular with compartment syndrome), b) causes a fall in haemoglobin level (Hb) of ≥2g/dL in a 24h period, or c) leads to transfusion of 2 or more units of whole blood or red blood cells (13).
* Suspected or confirmed bacterial endocarditis
* Ongoing or planned therapeutic anticoagulation for any other indication
* Platelet count <50,000/μL within the past 24 hours or Hb level <8g/dL
* Prothrombin time (PT) ≥2 seconds above the upper limit of age-appropriate local reference range within the past 24 hours
* Activated partial thromboplastin time (aPTT) ≥4 seconds above the upper limit of age-appropriate local reference range within the past 24 hours
* Fibrinogen <2.0 g/L
* Severe renal impairment (CrCl<30 mL/min) or acute kidney injury
* Use of dual antiplatelet therapy
* Pregnancy
* Unwillingness to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
mortality | Until patient is discharged or up to 4 weeks whichever comes first
  All cause mortality
occurrence of venous and/or arterial thrombosis | Until patient is discharged or up to 4 weeks whichever comes first
  clinical signs supported by radiological evidence of arterial thrombosis or venous thromboembolism (e.g. venous or arterial duplex and CT scan of the chest with pulmonary angiography)

SECONDARY OUTCOMES:
occurrence of Sepsis-induced coagulopathy | Until patient is discharged or up to 4 weeks whichever comes first
  calculation of sepsis induced coagulopathy (SIC) score
Occurrence of adult respiratory distress syndrome (ARDS) | Until patient is discharged or up to 4 weeks whichever comes first
  Calculation of partial pressure of arterial oxygen/ fraction of inspired oxygen (PaO2/ FIO2) ratio
Occurrence of sepsis | Until patient is discharged or up to 4 weeks whichever comes first
  Calculation of sequential organ failure (SOFA) score
ICU admission and need for mechanical ventilation | Until patient is discharged or up to 4 weeks whichever comes first
  occurrence of respiratory failure detected by arterial blood gases analysis

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Madkour, Principal Investigator — Ain Shams University, Faculty of Medicine
Locations (1):
- Faculty of Medicine Ain Shams University Research Institute- Clinical Research Center, Cairo, Non-US, Egypt

REFERENCES:
- [Derived] Flumignan RL, Civile VT, Tinoco JDS, Pascoal PI, Areias LL, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2022 Mar 4;3(3):CD013739. doi: 10.1002/14651858.CD013739.pub2. PMID 35244208